CLINICAL TRIAL: NCT02468089
Title: A Randomized Study to Compare the Efficacy of Carbepenem Versus Carbepenem Plus GM-CSF in Difficult To Treat Spontaneous Bacterial Peritonitis
Brief Title: To Compare the Efficacy of Carbepenem Versus Carbepenem Plus GM-CSF in Difficult To Treat Spontaneous Bacterial Peritonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-SBP-001
Record Dates: First submitted 2015-05-22; First posted 2015-06-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-01

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbepenem+albumin+GMCSF. (Experimental)
  Interventions: Drug: Carbepenem; Drug: Albumin; Drug: GMCSF (of Granulocyte-Monocyte Colony-Stimulating Factor) .
- Carbepenem+albumin (Active Comparator)
  Interventions: Drug: Carbepenem; Drug: Albumin

INTERVENTIONS:
Drug: Carbepenem
Drug: Albumin
Drug: GMCSF (of Granulocyte-Monocyte Colony-Stimulating Factor) .
  Arms: Carbepenem+albumin+GMCSF.

SUMMARY:
A Minimum of 150 consecutive patients of decompensated cirrhosis of any etiology, presenting to the Institute of Liver and Biliary Sciences hospital with a diagnosis of difficult to treat SBP will be included and randomized into two treatment groups.

Group A - Carbepenem+albumin Group B - Carbepenem+albumin+GMCSF.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years
2. Patients of decompensated liver cirrhosis who present with- Spontaneous bacterial peritonitis (Presence of more than 250 neutrophils per cc of ascetic fluid, in the absence of a surgical abdomen, in the presence of decompensated cirrhosis and portal hypertension) that is not responding to initial therapy- DTT-SBP:

   * Hospital acquired - New onset SBP (Spontaneous bacterial peritonitis) after 48 h of hospitalization.
   * Recurrent SBP - One or more prior episode(s) of SBP in year.
   * Antibiotic resistant - Resistance to 3rd Gen Cephalosporin in last 3 m.
   * Antibiotic non-response -Non-response to 3rd Gen Cephalosporin, sepsis on 3rd Gen Cephalosporin.

Exclusion Criteria:

1. < 18 years.
2. Advanced HCC (HepatoCellular Carcinoma)
3. Post liver transplant
4. HIV + ve, Immunosuppressive therapy
5. Pregnancy
6. Domiciliary treatment
7. No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Total no of patients cured from SBP (Spontaneous Bacterial Peritonitis) | 1 week

SECONDARY OUTCOMES:
Survival at week 2 | week 2
Survival at week 4 | week 4
Survival at week 12 | week 12
Total number of patients develop variceal bleed. | 1 week
Total number of patients develop non-SBP (Spontaneous Bacterial Peritonitis) infections within 1 wk of enrolment. | 1 week
Total number of patients develop HE (Hepatic Encephalopathy). | 1 week
Total number of patients develop AKI (Acute kidney Injury). | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Vikash Prakash, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India